CLINICAL TRIAL: NCT01484587
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CNTO 1959 Following a Single Subcutaneous Administration in Japanese Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics (What the Body Does to the Drug), and Pharmacodynamics (What the Drug Does to the Body) of CNTO 1959 Following a Single Subcutaneous (Under the Skin) Administration in Japanese Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR018646; CNTO1959PSO1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-09-02; First posted 2011-12-02 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Psoriasis
Keywords: Moderate to Severe Plaque-Type Psoriasis; Psoriasis; Plaque-type psoriasis; CNTO 1959; Japanese participants
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- 001 (Experimental)
  Interventions: Drug: CNTO 1959
- 002 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTO 1959 — CNTO 1959: type=range, unit=mg, number=10, 30, 100, 300, form=solution for injection, route=subcutaneous use, ascending dosing for 24 weeks
  Arms: 001
Drug: Placebo — Placebo: form=solution for injection, route=subcutaneous use, ascending dosing for 24 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to assess the safety and tolerability of CNTO 1959 following a single subcutaneous (SC, under the skin) dose administered to Japanese participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized (participants are assigned to treatment groups by chance), double-blind (participants and study personnel know what study agents are given), placebo-controlled (a placebo is a treatment identical in appearance to CNTO 1959 but does not contain active drug), single-dose study. The study will include 24 participants: 4 groups of at least 6 participants each. If it is decided that additional data are needed to define the safety and tolerability of CNTO 1959, an additional group may be enrolled. A given dose level may be repeated in newly enrolled participants, or a lower or intermediate dose may be administered based on preliminary data. The total duration of participation will be approximately 30 weeks, which includes a screening period of up to 6 weeks before the administration of study agent. Participant safety will be monitored. Ascending doses of 10, 30, 100, and 300 mg dose of CNTO 1959 and placebo will be administered as single SC injections; however, 2 SC injections may be required for the 300 mg dose level. Dosing will be performed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque-type psoriasis at least 6 months prior to screening (participants with concurrent psoriatic arthritis may be enrolled)
* Having plaque-type psoriasis covering at least 10% of total body surface area (BSA) at baseline
* Has a Psoriasis Area and Severity Index (PASI) score of 12 or greater at baseline
* Is a candidate for systemic phototherapy or systemic treatment of psoriasis (either new to treatment or having had previous treatment)
* Has at least 2 plaques suitable for repeat biopsy (Only participants who consent separately to participate in this assessment. Refusal to give consent for this component does not exclude an individual from participation in the clinical study).

Exclusion Criteria:

* Currently has non-plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular)
* Has current drug-induced psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (e.g., secondary infection occurred on bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), or open, draining, or infected skin wounds or ulcers
* Has a history of latent, or active or opportunistic systemic infection with pathogens including, but not limited to, Klebsiella pneumoniae, Cryptococcus neoformans, Candida albicans, Toxoplasma gondii, and Pneumocystis jiroveci prior to screening
* Has or has had a serious infection (e.g., sepsis, pneumonia or pyelonephritis), or have been hospitalized or received intravenous antibiotics for an infection during the 2 months prior to screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2013-04-11 (Actual); Study Completion 2013-04-11 (Actual)

PRIMARY OUTCOMES:
The number and type of adverse events | Up to 24 weeks
Change in clinical laboratory values | Up to 24 weeks
Electrocardiogram | Up to 24 weeks
Changes or abnormalities in body systems | Up to 24 weeks
Axillary temperature | Up to 24 weeks
Pulse rate | Up to 24 weeks
Blood pressure | Up to 24 weeks

SECONDARY OUTCOMES:
Blood levels of CNTO 1959 | Up to 24 weeks
Antibodies to CNTO 1959 | Up to 24 weeks
Psoriasis Area and Severity Index (PASI) | Up to 24 weeks
  The PASI produces a numeric score that can range from 0 (no involvement) to 72 (90% to 100% involvement).
Physician's Global Assessment (PGA) | Up to 24 weeks
  Assessment of the patient's psoriasis status according to the following categories: induration, erythema, and scaling

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Sapporo, Japan

REFERENCES:
- See also: Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CNTO 1959 following a Single Subcutaneous Administration in Japanese Subjects With Moderate to Severe Plaque Psoriasis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3368&filename=CR108646_CSR.pdf